CLINICAL TRIAL: NCT01544959
Title: The Impact on Postoperative Pain of Substituting Opioids by Beta Blockers for Peroperative Hemodynamic Control in Patients Undergoing Mastectomy
Brief Title: Postoperative Analgesia Impact of Narcotic Free Anesthesia
Acronym: PAINFree
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Etienne de Medicis, Doctor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRC-09-174; CAS-008-2010 (Other Grant/Funding Number: CAS/Vitaid Award)
Record Dates: First submitted 2010-09-09; First posted 2012-03-06 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative; Breast Cancer; Postoperative Nausea and Vomiting
Keywords: Narcotic; Opioid; betablocking drug; postoperative pain; postoperative nausea and vomiting; breast cancer; hyperalgesia; cancer recurrence; anesthesia; mastectomy; chronic postsurgical pain syndrome; acute postoperative pain; postmastectomy pain syndrome; pain; ambulatory surgery
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms; Postoperative Nausea and Vomiting; Hyperalgesia; Pain | interventions — Fentanyl; Adrenergic beta-Antagonists; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl (Active Comparator)
  Interventions: Drug: fentanyl
- beta-blocker (Experimental): Instead of narcotics (fentanyl), esmolol and lopressor are being used for hemodynamic control
  Interventions: Drug: beta-blocker (esmolol, metropolol)

INTERVENTIONS:
Drug: fentanyl — Use of esmolol and metoprolol compared to use of fentanyl for hemodynamic control during general anesthesia. At induction, fentanyl (2 mcg/kg) is replaced by esmolol (1 mg/kg). During the case, with a standardised anesthesia, response to surgical stimulation will be medicated either by fentanyl (50 mcg aliquot) or metropolol (2.5 mg), for a maximum of 6 doses. After this, fentanyl will be given unblindly.
  Arms: fentanyl
Drug: beta-blocker (esmolol, metropolol) — esmolol is used at induction and lopressor during surgery instead of fentanyl in response to surgical stimulation.
  Arms: beta-blocker

SUMMARY:
The first hypothesis of the study is that substituting fentanyl by esmolol and metoprolol during general anesthesia for patients undergoing mastectomy will result in less pain and less narcotic consumption in the recovery room. The investigators will also verify the impact of that substitution on nausea and vomiting, on the time spent in the recovery room and on chronic postsurgical pain (3 and 6 months).

Finally, the investigators will see the impact on breast cancer recurrence 5 years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* 18 to 65 years old
* ASA 1 or 2
* First breast surgery
* Unilateral breast cancer
* Partial mastectomy or radical modified mastectomy ± axillary dissection

Exclusion Criteria:

* Allergy or contrindication to any medication figuring in the protocol or to Aspirin
* Patient taking betablocking drug drug or lanoxin or calcic channels blocking drug
* Narcotic consumption in the past month of 10 mg/day of morphine equivalent
* Chronic pain
* Moderate to severe asthma
* BMI of more than 40
* Diabetes
* Chronic renal or hepatic faiure
* Heart failure
* Anticipated difficult airway
* High grade heart block or bifascicular block
* Mental retardation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Postoperative consumption of narcotic in recovery room | Immediately after surgery

SECONDARY OUTCOMES:
Pain level in recovery room | immediately after surgery
Occurence of nausea and vomiting in the recovery room | immediately after surgery
Time spent in recovery room | immediately after surgery
Chronic post-surgical pain | 3 and 6 months
Reccurence of breast cancer | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Etienne de Medicis, MD MSc, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada